CLINICAL TRIAL: NCT04819893
Title: Study of the Involvement of Fatty Acids in Retinopathy of Prematurity: Relationship Between Retinopathy of Prematurity and the Rate of Expression of Transplacental Fatty Acid Receptors.
Acronym: OMEGAROP 2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: CREUZOT-GARCHER 2020-1
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prematurity; Retinopathy
MeSH Terms: conditions — Premature Birth; Retinal Diseases | interventions — Cordocentesis; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women giving birth prematurely: Delivery before 29 WA
  Interventions: Biological: Maternal blood sampling; Biological: Umbilical cord blood sampling; Biological: Placenta sampling; Other: Data collection
- Women giving birth at term: Childbirth between 39WA and 31WA+6 days
  Interventions: Biological: Maternal blood sampling; Biological: Umbilical cord blood sampling; Biological: Placenta sampling

INTERVENTIONS:
Biological: Maternal blood sampling — 5 mL sample of venous blood on arrival at the maternity ward in accordance with standard protocols
Biological: Umbilical cord blood sampling — 0.5mL sample from the umbilical cord after childbirth standard protocols
Biological: Placenta sampling — Sampling of 3 cotyledons by cutting across the thickness of the placenta
Other: Data collection — Newborn, Maternal and Premature Retinopathy Screening Data Collection
  Groups: Women giving birth prematurely

SUMMARY:
The development of the retinal vascular network is completed during the third trimester of pregnancy and and the first 15 days of life of the newborn. This late maturation can be problematic in cases of preterm births and result in immature retinal vascularization, known as retinopathy of prematurity (ROP). Among the various factors influencing retinal vascular development, the tissue content of omega-3 polyunsaturated fatty acids (PUFAs) appears to be a crucial element. In a previous project, OMEGA-ROP, we showed a difference in the blood bioavailability of omega-3 PUFAs in infants born at less than 28 weeks of amenorrhea who develop ROP compared to healthy newborns with no retinopathy. This study also showed that mothers experienced variations in the blood levels of omega-3 PUFAs that were contrary to the types of variations observed in their children. This suggests a sequestration of omega-3 PUFAs in the mothers of children who will develop ROP. This new project aims to better understand the underlying molecular mechanisms by studying the expression levels of placental fatty acid receptors in relation to the development of ROP in newborns.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers giving birth to premature babies less than 29 weeks of amenorrhea (WA), after obtaining their non-opposition.
2. Mothers giving birth at term between 39 and 41WA+6 days, after obtaining their non-opposition.
3. ≥18 years
4. Mothers not under legal protection

Exclusion Criteria:

1. Mothers giving birth between 29WA and 38WA+6 days
2. Mothers in critical condition.
3. Person not affiliated to national health insurance
4. For full-term mothers: patient presenting or having presented a health condition that affected a previous pregnancy (vascular such as pregnant hypertension, preeclampsia; gestational diabetes; intrauterine growth retardation, maternal infection during pregnancy such as toxoplasmosis, cytomegalovirus, rubella, measles, chickenpox).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Women giving birth at term or prematurely
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Estimation of the linear correlation coefficient between placental fatty acid receptor expression rate and term of delivery | 16 weeks maximum after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carre C, Acar N, Daruich A, Gregoire S, Martine L, Buteau B, Aho S, Eid P, Arnould L, Bron AM, Driessen M, Kermorvant E, Simon E, Creuzot-Garcher C, Gabrielle PH. Study protocol of OmegaROP-2 prospective study: expression of placental fatty acid receptors in preterm newborns with retinopathy of prematurity. BMC Ophthalmol. 2023 Oct 6;23(1):404. doi: 10.1186/s12886-023-03156-0. PMID 37803473